CLINICAL TRIAL: NCT05538819
Title: The Effects of Glimepiride in Patients With Type 2 Diabetes and Chronic Heart Failure
Acronym: EGPT2D&CHF
Status: Completed | Type: Observational
Sponsor: Dao Wen Wang (Other)
Collaborators: Shanghai Institute of Materia Medica, Chinese Academy of Sciences (Other)
Responsible Party: Sponsor-Investigator, Dao Wen Wang, Prof., Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-T2D&CHF-Glimepiride
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic Heart Failure; Type 2 Diabetes; Cardiovascular Mortality; Cohort Study
Keywords: glimepiride; type 2 diabetes; chronic heart failure; cardiovascular mortality
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glimepiride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Glimepiride group: 509 patients aged >18 years with T2D and CHF had continuous glimepiride use (1-4 mg/day).
  Interventions: Drug: Glimepiride
- Non-glimepiride group: 509 patients aged >18 years with T2D and CHF had no glimepiride use.

INTERVENTIONS:
Drug: Glimepiride — Glimepiride 1-4 mg/day
  Other Names: Amaryl
  Groups: Glimepiride group

SUMMARY:
Thirty years ago, Dzau and Braunwald introduced the concept of a continuum of cardiovascular diseases and defined them as a series of events caused by numerous related and unrelated risk factors, thus developing to end-stage heart disease through many pathophysiological pathways and processes. Owing to treatment concept changes and the urgency of investigating T2D combined with CHF, SUs are being re-evaluated, of which glimepiride is undoubtedly the most promising.

DETAILED DESCRIPTION:
Since the first sulfonylurea (SU; tolbutamide) was commercially launched in Germany in 1956, SUs, as the oldest oral hypoglycemic drugs, have been developed for three generations and are commonly used for patients with T2D. In 2008, the US Food and Drug Administration and European Drug Administration required cardiovascular safety certification for all hypoglycemic drugs, resulting in increased related clinical trials. Currently, data on the relationship between SUs and cardiovascular outcomes are limited, and the cardiovascular effects remain controversial in observational studies. Third-generation SUs, such as glimepiride, are widely used for treating T2D because of their definite hypoglycemic efficacy, relatively low risk of hypoglycemia, convenient daily use, and low price. Glimepiride has good cardiovascular safety according to randomized controlled trials (RCTs). The proportion of SUs used in patients with heart failure is as high as 60.4%. Although some studies have shown that SUs are neutral in terms of hospitalization rates and adverse cardiovascular events in patients with CHF, no standard RCT of glimepiride has been conducted to study its effect on the prognosis of patients with T2D and confirmed CHF. Glimepiride inhibits soluble epoxide hydrolase (sEH), thus reducing epoxyeicosatrienoic acid (EET) degradation . Increased EET production exerts protective effects on the heart, indicating the potential cardiovascular effect of glimepiride.

This retrospective cohort study aimed to evaluate the effects of glimepiride on the clinical outcomes of patients with T2D and CHF and provide theoretical evidence for the clinical application of glimepiride in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure (>6 months duration, according to 2021 ESC Guidelines for the Diagnosis and Treatment of Acute and Chronic Heart Failure)
* Reduced ejection fraction defined as LVEF < 50%
* N-terminal pro-brain natriuretic peptide (NT-proBNP) level: >125 pg/mL
* NYHA-class II/III/IV with stable symptoms for at least the past 3 months
* Type 2 diabetes (according to the Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2022)

Exclusion Criteria:

* Those who did not meet the diagnostic criteria
* Lacked echocardiographic and NT-proBNP data
* Used sulfonylureas other than glimepiride were excluded

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: According to continuous glimepiride use, the patients were divided into glimepiride and non-glimepiride groups. A 1:1 propensity score matching (PSM) analysis was used to balance the confounding factors between the glimepiride treatment and clinical outcomes. The PSM cohort (509:509) was followed up using a telephone questionnaire directly or at an outpatient clinic at our cardiac center. The follow-up deadline was July 1, 2022. According to the follow-up results, the glimepiride group was subdivided into high-dose (2-4 mg/day) and low-dose (1 mg/day) groups.
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Cardiovascular mortality | 5 years
  Numbers and dates of death due to cardiovascular diseases in each group
Hospitalizations and emergency visits for heart failure | 5 years
  Numbers and dates of hospitalizations and emergency for heart failure

SECONDARY OUTCOMES:
All-cause mortality | 5 years
  Numbers and dates of death in each group
Hospitalizations for acute myocardial infarction or stroke | 5 years
  Numbers and dates of hospitalizations for acute myocardial infarction or stroke

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
We are working hard to have IPD sharing plan and are willing to share it with other researchers.

REFERENCES:
- [Derived] He W, Yuan G, Han Y, Yan Y, Li G, Zhao C, Shen J, Jiang X, Chen C, Ni L, Wang DW. Glimepiride Use is Associated with Reduced Cardiovascular Mortality in Patients with Type 2 Diabetes and Chronic Heart Failure: A Prospective Cohort Study. Eur J Prev Cardiol. 2022 Dec 27:zwac312. doi: 10.1093/eurjpc/zwac312. Online ahead of print. PMID 36573717